CLINICAL TRIAL: NCT03665922
Title: Biomarkers of Sulforaphane/Broccoli Sprout Extract in Prostate Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Bruce Jacobs, Univ of P. Physicians Faculty, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: STUDY19050340; R01CA225716 (NIH)
Record Dates: First submitted 2018-09-05; First posted 2018-09-11 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Prostate Cancer
Keywords: prostatectomy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — microcrystalline cellulose

STUDY DESIGN:
Intervention Model Description: Double-blind randomized placebo controlled design
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BroccoMax® (Experimental): Following randomization, subjects will begin to take four BroccoMax® tablets in the morning with breakfast and four tablets in the evening with dinner. The eight BroccoMax® tablets will provide a daily internal dose of 64 mg of SFN.
  Interventions: Dietary Supplement: BroccoMax®
- Placebo (Placebo Comparator): Following randomization, subjects will begin to take four placebo tablets in the morning with breakfast and four tablets in the evening with dinner.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: BroccoMax® — Nutraceutical neoadjuvant
  Arms: BroccoMax®
Other: Placebo — control
  Other Names: Microcrystalline cellulose
  Arms: Placebo

SUMMARY:
This study will test whether oral intake of a dietary supplement called BroccoMax®, which is a special blend of broccoli extract containing a chemical called sulforaphane (hereafter abbreviated as SFN), may result in changes in chemicals that feed prostate cancer. BroccoMax® is available over the counter.

DETAILED DESCRIPTION:
Eligible subjects will be randomly assigned to either BroccoMax® or placebo arm with a 1:1 randomization. Each subject will be given BroccoMax® equivalent to 4 weeks supply. Following randomization, subjects will begin to take four study tablets (BroccoMax® or placebo) in the morning with breakfast and four tablets in the evening with dinner. The eight BroccoMax® tablets will provide a daily internal dose of 64 mg of SFN.

Baseline evaluation will be 28 days before scheduled prostatectomy, the same day of study drug dispensation, and will include.

1. Data collection on patient's medical history (which includes age, cancer history, review of medications, food intolerances and food habits), and concomitant medications.
2. Physical exam including height and weight measurements.
3. Blood (approximately 15 mL) will be collected in Serum Separator Tube-tiger tubes (SST)for determination of SFN and its metabolite levels and for biomarker analyses.
4. Spot urine collection (15 mL) for measuring SFN and its metabolite levels.
5. Four-week supply of study drug (BroccoMax® or Placebo) dispensation

Day 28 ± 3 days (End of study evaluation)

1. Physical exam including height and weight measurements
2. Blood (approximately 15 mL) will be collected in SST-tiger tubes for determination of SFN and its metabolite levels and for biomarker analyses.
3. Spot urine collection (15 mL) for measuring SFN and its metabolite levels.
4. Adverse event assessment.
5. A portion of the prostate tumor after surgical resection will be fresh frozen in liquid nitrogen.
6. After pathological assessment is complete, tumor blocks or slides (6 or more) will be requested by the clinical research coordinator from the Health Sciences Tissue Bank of the University of Pittsburgh for biomarker analyses.

Post-Treatment Follow-Up All study participants will have routine follow-up as determined by their treating urologist and/ or medical oncologist. This usually occurs 6 ± 2 weeks post-surgery and every 3 months thereafter. These are considered standard of care visits. The patient chart will be reviewed for their history and physical findings at these visits.

ELIGIBILITY:
Inclusion Criteria:

1. Men ≥ 18 years of age scheduled to undergo radical prostatectomy as standard of care for a diagnosis of prostate adenocarcinoma.
2. Subjects willing to take oral placebo or BroccoMax® pills (4 capsules twice daily after breakfast and dinner) on a daily basis for 4 weeks prior to prostatectomy. Subjects have the ability to swallow BroccoMax® or placebo pills.
3. Subjects in good health per investigator evaluation with liver enzyme and blood count values within the following ranges:

   White blood cells ≥ 3,000/mL Total bilirubin ≤ 1.5 x Upper Limits of Normal (ULN) Aspartate Aminotransferase (AST (SGOT))/ Alanine Aminotransferase (ALT (SGPT)) ≤ 2.5 x ULN Blood Urea Nitrogen (BUN) and serum creatinine ≤ 1.5 x ULN
4. Subjects willing to abstain from dietary sources of glucosinolates and isothiocyanates (see Appendix) for the duration of the study (4 weeks)
5. Subjects must be fully informed of the investigational nature of this study and must sign a written informed consent in accordance within institutional and regulatory guidelines

Exclusion Criteria:

1. Subjects ineligible to undergo prostatectomy due to co-morbidities.
2. Subjects with a second malignancy or any other cancer at least 3 years following definitive treatment with no evidence of disease, except for adequately treated basal cell or squamous cell skin cancer.
3. Subjects with malabsorption issues or gastrointestinal ailments than can interfere with the ability to adequately absorb SFN.
4. Subjects with prior or concurrent androgen deprivation therapy with Luteinizing hormone-releasing hormone (LHRH) agonist or antagonists
5. Subjects taking any other investigational agent, dietary supplement or herbal supplement or participating in clinical studies involving investigational agents
6. Subjects with clinically significant comorbid diseases including active infection, uncontrolled angina, New York Heart Assoc. (NYHA) class III or IV heart failure, uncontrolled or uncontrollable hypertension, severe diabetes with complications, chronic liver disease.
7. Subjects with prior history of known intolerance or allergic reactions attributed to cruciferous vegetables or specific fillers used in the placebo.

Ages: 18 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Palmitic Acid Reduction | 4 weeks
  Change in serum levels of palmitic acid (the primary free fatty acid) in subjects treated with BroccoMax® compared to placebo.

SECONDARY OUTCOMES:
Evaluation of safety of BroccoMax® (side effects or adverse events) | 2 months
  Assessing any side effects or adverse events that could be associated with the oral intake of BroccoMax®
Serum SFN levels | 4 weeks
  Compare the levels of SFN and its metabolites in serum at day 14 and week 4 to baseline
Urine SFN levels | 4 weeks
  Compare the levels of SFN and its metabolites in urine at day 14 and week 4 to baseline.
Prostate adenocarcinoma SFN level | Week 4
  Evaluate the SFN and its metabolites in the prostate/ prostate adenocarcinoma tissue.
Mean proliferative index (Ki-67) and apoptotic marker (TUNEL) in prostate adenocarcinoma sections | Week 4
  Evaluate the biomarkers of the collected tissue.
Evaluation of Prostate adenocarcinoma tissue by immunohistochemistry. | Week 4
  Prostate adenocarcinoma expression of acetyl-Coenzyme A carboxylase 1 (ACC1), fatty acid synthase (FASN), carnitine palmitoyltransferase1A (CPT1A), androgen receptor (AR), phosphatase and tensin homolog (PTEN), sterol regulatory binding protein 1 (SREBP-1) and c-Myc by immunohistochemistry (IHC)
Evaluation of serum levels of fatty acid metabolism intermediates. | Weeks 2 and 4.
  Evaluate Serum levels of Acetyl-Coenzyme A, Malonyl-Coenzyme A, total phospholipids, adenosine triphosphate (ATP), and global lipidemic
Evaluation of prostate adenocarcinoma levels of fatty acid metabolism intermediates | Week 4
  Evaluate prostate adenocarcinoma levels of Acetyl-Coenzyme A, Malonyl-Coenzyme A, total phospholipids, ATP, and global lipidemic

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Jacobs, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- Shadyside Urology, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Siegel RL, Miller KD, Jemal A. Cancer Statistics, 2017. CA Cancer J Clin. 2017 Jan;67(1):7-30. doi: 10.3322/caac.21387. Epub 2017 Jan 5. PMID 28055103
- [Background] Key T. Risk factors for prostate cancer. Cancer Surv. 1995;23:63-77. PMID 7621474
- [Background] Roobol MJ, Carlsson SV. Risk stratification in prostate cancer screening. Nat Rev Urol. 2013 Jan;10(1):38-48. doi: 10.1038/nrurol.2012.225. Epub 2012 Dec 18. PMID 23247693
- [Background] Drudge-Coates L, Turner B. Prostate cancer overview. Part 2: metastatic prostate cancer. Br J Nurs. 2012 Oct 11-24;21(18):S23-4, S26-8. PMID 23123814
- [Background] Mitchell T, Neal DE. The genomic evolution of human prostate cancer. Br J Cancer. 2015 Jul 14;113(2):193-8. doi: 10.1038/bjc.2015.234. Epub 2015 Jun 30. PMID 26125442
- [Background] Ju J, Picinich SC, Yang Z, Zhao Y, Suh N, Kong AN, Yang CS. Cancer-preventive activities of tocopherols and tocotrienols. Carcinogenesis. 2010 Apr;31(4):533-42. doi: 10.1093/carcin/bgp205. Epub 2009 Sep 11. PMID 19748925
- [Background] Lee KW, Bode AM, Dong Z. Molecular targets of phytochemicals for cancer prevention. Nat Rev Cancer. 2011 Mar;11(3):211-8. doi: 10.1038/nrc3017. Epub 2011 Feb 10. PMID 21326325
- [Background] Saha A, Blando J, Silver E, Beltran L, Sessler J, DiGiovanni J. 6-Shogaol from dried ginger inhibits growth of prostate cancer cells both in vitro and in vivo through inhibition of STAT3 and NF-kappaB signaling. Cancer Prev Res (Phila). 2014 Jun;7(6):627-38. doi: 10.1158/1940-6207.CAPR-13-0420. Epub 2014 Apr 1. PMID 24691500
- [Background] Kallifatidis G, Hoy JJ, Lokeshwar BL. Bioactive natural products for chemoprevention and treatment of castration-resistant prostate cancer. Semin Cancer Biol. 2016 Oct;40-41:160-169. doi: 10.1016/j.semcancer.2016.06.003. Epub 2016 Jun 28. PMID 27370570
- [Background] Thompson IM, Goodman PJ, Tangen CM, Lucia MS, Miller GJ, Ford LG, Lieber MM, Cespedes RD, Atkins JN, Lippman SM, Carlin SM, Ryan A, Szczepanek CM, Crowley JJ, Coltman CA Jr. The influence of finasteride on the development of prostate cancer. N Engl J Med. 2003 Jul 17;349(3):215-24. doi: 10.1056/NEJMoa030660. Epub 2003 Jun 24. PMID 12824459